CLINICAL TRIAL: NCT06291753
Title: Characteristics and Tumor Staging Proposal for Primary Malignant Melanoma of the
Brief Title: Characteristics and Tumor Staging Proposal for Primary Malignant Melanoma of the Esophagus
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Weijie Ye, Principal Investigator, Sun Yat-sen University
Other Study IDs: SL-B2023-478-01
Record Dates: First submitted 2024-02-18; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Primary Malignant Melanoma of the Esophagus
Keywords: cancer of esophagus, melanoma, overall survival, surgery, tumor staging
MeSH Terms: conditions — Esophageal Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Primary malignant melanoma of the esophagus (PMME) is a malignant tumor originating from esophageal melanocytes with a poor prognosis. No international clinical guidelines or tumor staging systems have been proposed for PMME. This study aimed to analyze the clinical characteristics and treatment outcomes of patients with PMME and propose a tumor staging system in PMME.

Materials and Methods: The clinical characteristics of 25 patients with PMME at our cancer center were summarized, and 21 patients were enrolled in a pooled analysis with 162 cases (extracted from 74 eligible articles in PubMed) for further survival analysis and proposal of PMME tumor staging.

DETAILED DESCRIPTION:
Introduction Melanoma is a malignant tumor that originates from chromatophores. Primary malignant melanoma of the esophagus (PMME) grows from esophageal melanocytes, accounting for 3.8% of mucosal melanoma and 0.1%~0.2% of esophageal malignant tumors.PMME is highly malignant with a 5-year overall survival (OS) less than 5%. Typical PMME cases in endoscopy or surgical specimens usually show a well-circumscribed, elevated, and black-pigmented tumor. Some "amelanotic melanoma" cases lack melanin pigmentation in PMME. Regarding this disease, melanin-producing melanocytes exhibit various growth patterns and progression, irregular, spindle-shaped, and epithelioid cell structures. Solid tumor cells proliferation and nests formation are commonly observed in pathological slides. Baur reported the first case of malignant esophageal melanoma in 1906; however, Pava discovered the typical melanocytes in the esophageal epithelium in 1963, which was considered a primary malignant esophageal tumor. In 1989, Pradhan added the most common PMME sites, including its histological and cytological characteristics. Studies show that esophageal melanoma is similar to mucosal melanoma and presents very different features from skin, marginal or basal melanoma. PMME diagnosis usually depends on the following criteria: (1) a typical histological melanoma pattern, with melanin granules inside the tumor cells. (2) origin in an area of junctional activity in squamous epithelium. Moreover, positive immunohistochemical staining for S-100, HMB45, Melan-A, and CK (AE1/AE3) can significantly contribute to the confirmation of a definitive PMME diagnosis.

Owing to the rarity of PMME, with ≤ 500 cases currently reported , few researchers have focused on effective treatments and drug selection for postoperative adjuvant therapy. As only a few cases and unique biological characteristics of PMME exist, tumor staging, such as esophageal squamous cell carcinoma (ESCC) or esophageal adenocarcinoma (EAC), is unsuitable for guiding PMME treatment and prognosis. No specific international clinical guidelines or standard tumor, node, metastasis (TNM) staging systems exist for PMME. Surgical resection remains the most effective method for treating PMME, and patients who underwent surgery without adjuvant or neoadjuvant therapy had median OS ranging from 8.0 to 34.5 months. Owing to the low PMME incidence rate, large-scale prospective research is almost impossible to conduct to confirm the effectiveness and courses of chemotherapeutics for PMME. Presently, PMME treatment is still based on the guidelines for cutaneous melanoma and other pathological esophageal cancer types. Therefore, further studies are required to explore the PMME treatment. This study aimed to analyze the clinical characteristics and treatment outcomes of patients with PMME and propose a tumor staging system for PMME.

Material and Methods Patient selection and recurrence monitoring at our cancer center Detailed patient data were collected from the database of the Sun Yat-sen University Cancer Center, and the PMME diagnosis was confirmed through the pathological diagnosis of the surgical specimen and immunohistochemical staining. The pathological stages of the patients were reassessed following the 8th edition of the Union for International Cancer Control (UICC) and American Joint Committee on Cancer (AJCC) TNM classification system. Follow-up was conducted via telephone to record the living status and time of death.Survival analysis for pooled data and strategy for cancer stage reorganization.

Survival analysis for pooled data and strategy for cancer stage reorganization To verify the findings based on survival analysis of patients at the Sun Yat-sen University Cancer Center, we collected eligible original data from PubMed for further survival analysis and proposed a new tumor staging system for PMME. Univariate and multivariate Cox regression analysis were used to analyze the independent prognostic factors. OS was used instead of melanoma-specific survival to describe the actual situation in this study. Melanoma and esophagus and esophagogastric junction staging in 8th AJCC edition were used as references. All TNM staging extracted from the screened studies was reassessed in 8th AJCC edition of esophagus and esophagogastric junction staging. Based on the independent prognostic factors analyzed, pathological PMME tumor staging was proposed. Overall, the purpose of tumor staging was to group cancer features to reflect the decrease in OS in the increasing staging group (monotonicity), differences in OS between groups (uniqueness), and similar OS within groups (homogeneity).

Literature research Literature on PMME published between March 1950 and August 2023 was searched on PubMed using the keyword "Primary malignant melanoma of esophagus." The search date was August 28, 2023. The following selection criteria were used: 1) primary malignant melanoma of esophagus confirmed via biopsy; autopsy; endoscopic mucosal resection and dissection and specimen in pathologic diagnosis; 2) patients who had been followed up for ≥6 months or reached endpoint event; 3) cases reported in the English literature. The exclusion criteria were as follows: 1) patients with primary malignant melanoma of esophagus and other esophageal tumors, 2) patients without a clear TNM stage or who could not be reassessed using 8th AJCC edition of esophagus and esophagogastric junction cancer staging manual. The information from each patient was carefully reviewed by two authors and any repeated patients were excluded. The information on the patients collected included the location of the tumor; radiotherapy and chemotherapy after surgery; and tumor recurrence or progression. The pTNM stages were reassessed in AJCC 8th edition of esophagus and esophagogastric junction cancer staging manual.

ELIGIBILITY:
Inclusion Criteria:

1. primary malignant melanoma of esophagus confirmed via biopsy; autopsy; endoscopic mucosal resection and dissection and specimen in pathologic diagnosis
2. patients who had been followed up for ≥6 months or reached endpoint event

Exclusion Criteria:

1. patients with primary malignant melanoma of esophagus and other esophageal tumors
2. patients without a clear TNM stage or who could not be reassessed using 8th AJCC edition of esophagus and esophagogastric junction cancer staging manual

Ages: 23 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Detailed patient data were collected from the database of the Sun Yat-sen University Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-02-18 (Actual); Study Completion 2024-02-18 (Actual)

PRIMARY OUTCOMES:
Overall Survival(OS) | From date of disease diagnosis until the date of death from any cause, assessed up to 170 months
  Overall Survival (OS) is a term used in oncology and clinical trials to refer to the length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive.
Disease-free survival (DFS) | From the date of the initial treatments in Sun Yat-sen University Cancer Center to the recurrence of the disease or death due to any cause, assessed up to 170 months
  Disease-free survival (DFS) is defined as the time from randomization to recurrence of tumor or death, and it is typically used in the adjuvant treatment setting.

CONTACTS AND LOCATIONS:
Locations (1):
- Qianwen Liu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No